CLINICAL TRIAL: NCT04193774
Title: Optimization of Sampling for Molecular Microbial Research on Ocular Surface Samples and Building a Framework for Comparing Current Sequencing Results Using Different Extraction Protocols.
Brief Title: Optimization of Sampling and Processing of Samples for Molecular Microbial Research on Ocular Surface Samples
Acronym: EPSO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: S62672
Record Dates: First submitted 2019-12-04; First posted 2019-12-10 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-06

CONDITIONS: Microbiota; Ocular Surface
Keywords: Ocular surface microbiome; Anesthesia; Extraction protocol
MeSH Terms: interventions — benoxinate; Ophthalmic Solutions; Anesthetics; Lubricant Eye Drops

STUDY DESIGN:
Intervention Model Description: When the patient is under general anesthesia for another reason, he or she receives a drop of artificial tears in one eye and a drop of anesthetic in the other eye in a randomized way.
Who Masked: Care Provider, Investigator
Masking Description: The nurse application the drops receives a closed envelope wherein the information about which eye receives what type of drop is included. The executor is blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drop of artificial tears (Placebo Comparator): A drop op Thealoz duo
  Interventions: Diagnostic Test: Conjunctival swab; Drug: artificial tears
- Drop op anesthetic (Active Comparator): A drop of oxybuprocaïne
  Interventions: Diagnostic Test: Conjunctival swab; Drug: Oxybuprocaine Hydrochloride 0.4% Eye Drops

INTERVENTIONS:
Diagnostic Test: Conjunctival swab — Swab of the conjunctival fornices of both eyes
Drug: Oxybuprocaine Hydrochloride 0.4% Eye Drops — One drop of topical anesthesia in one eye
  Other Names: anesthetic
  Arms: Drop op anesthetic
Drug: artificial tears — One drop of artificial tears in the other eye
  Other Names: Thealoz duo
  Arms: Drop of artificial tears

SUMMARY:
The use of anesthetics and the processing of the retrieved samples are major confounding factors that influence the results of microbiome research.

DETAILED DESCRIPTION:
The use of anesthetics is subject of discussion in ocular surface microbiome research. One publication showed a significant lower alpha diversity when using an anesthetic. However, the diluting effect of the anesthetic drop itself was not accounted for. On the other hand, using anesthetics will enable patients to tolerate sampling better and this might allow better sampling. To analyze the effect of anesthetic drops on the composition of the ocular surface microbiome, we sampled volunteers undergoing general anesthesia. By using artificial tears as a control, we aimed at accounting for the diluting effect of the anesthetic. By using volunteers under general anesthesia, we wanted to assure similar pressure with or without topical anesthesia since the executor was not influenced by the patient's reaction.

Furthermore, the effect of different extraction protocols on sequencing results will be assessed by sampling different volunteers in both eyes on non consecutive days.

ELIGIBILITY:
Inclusion Criteria:

* Willing to undergo sampling of the conjunctiva
* Fluent in written and verbal Dutch
* Capable of giving informed consent

Exclusion Criteria:

* Allergy to oxybuprocaine
* Medication usage in one eye only

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-08-19 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Difference in richness of the microbial flora measured as operational taxonomic units | 5 minutes per sampling session
  The difference in richness and evenness of distribution of the microbial flora of samples retrieved after a drop of topical anesthesia versus samples retrieved after a drop of artificial tears.
Difference in evenness of distribution of the microbial flora measured as operational taxonomic units | 5 minutes per sampling session
  The effect of the different microbial DNA extraction protocols on the richness and evenness of distribution of the microbial flora of the ocular surface will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Heleen Delbeke, MD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- University Hospitals Leuven, Department of Ophthalmology, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-01): https://cdn.clinicaltrials.gov/large-docs/74/NCT04193774/Prot_SAP_000.pdf